CLINICAL TRIAL: NCT05545631
Title: Microbiome and Transcriptome Predicts Pregnancy Outcomes Undergoing Frozen Embryo Transfer: A Multicenter Prospective Observational Study
Brief Title: Frozen Embryo Transfer Pregnancy Outcomes Prediction by Microbiome and Transcriptome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shengjing Hospital (Other)
Collaborators: Beijing Institutes of Life Science, Chinese Academy of Sciences (Unknown)
Responsible Party: Principal Investigator, Xiuxia Wang, Principal Investigator, Shengjing Hospital
Other Study IDs: Shengjing Hospital 1
Record Dates: First submitted 2022-09-15; First posted 2022-09-19 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Infertility; Microbiome
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Conception positive: serum human chorionic gonadotropin ≥10 mIU/mL
  Interventions: Other: no intervention
- Conception negative: serum human chorionic gonadotropin <10 mIU/mL
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention in this study

SUMMARY:
This study intends to explore the correlation between cervical microbiome, gut microbiome, transcriptome and pregnancy outcomes of frozen embryo transfer patients through a multicenter prospective observational study, and to explore the predictive value of microbiome on pregnancy outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Infertile women receiving assisted reproductive technology treatment, preparing for frozen embryo transfer cycle;
2. Female age: 20-45 years old;
3. Single frozen-thawed blastocyst Transferred
4. Endometrial thickness ≥7mm on the day of luteal transformation
5. Written informed consent.

Exclusion Criteria:

1. Women who have pathologies or malformations that affect the pregnancy outcome:genital malformations, intrauterine adhesions, uterine fibroids (>4 cm in diameter or compressing endometrial line), adenomyosis, endometrial polyps; untreated tubal pleura Presence of autoimmune disease;
2. Untreated hyperprolactinemia, thyroid disease, adrenal disease
3. Antibiotic use within the past 7 days;
4. Current or recent (within 3 months) drug abuse, including alcohol and tobacco;
5. Refused or unable to comply with protocol requirements;
6. Participation in any experimental drug study within 60 days prior to screening.

Ages: 20 Years to 45 Years | Sex: Female
Age Groups: Adult
Study Population: Patients attending Center of Reproductive Medicine
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Concentration of serum human chorionic gonadotropin ≥10 mIU/mL | 09.01.2022 to 09.01.2024
  Conception

SECONDARY OUTCOMES:
Clinical pregnancy | 09.01.2022 to 09.01.2024
  detection of a gestational sac in the uterine cavity 3 weeks after conception

CONTACTS AND LOCATIONS:
Overall Officials: Xiuxia Wang, Doctor, Principal Investigator — Center of Reproductive Medicine, Shengjing Hospital of China Medical University; Sufen Cai, Doctor, Principal Investigator — Reproductive and Genetic Hospital of CITIC-Xiangya
Locations (1):
- Xiuxia Wang, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No